CLINICAL TRIAL: NCT03473912
Title: Rheumatologic Biobank for Clinical and Basic Research: Isolation, Extraction and Storage of Protein, DNA and RNA Extracted From Tissues of Patients With Rheumatoid Diseases
Brief Title: Meir Medical Center Rheumatologic Biobank
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC17-0116CTIL
Record Dates: First submitted 2017-09-10; First posted 2018-03-22 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis; Lupus Erythematosus, Systemic; Systemic Sclerosis; IgG4-related Disease; Sjogren's Syndrome
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Immunoglobulin G4-Related Disease; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — blood, synovial fluid and skin biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RA patients: before or after medication
- Systemic sclerosis patients: before or after medication
- IgG4 RD patients: before or after medication
- Lupus patients: before or after medication

SUMMARY:
Serum, synovial fluid and skin biopsies from patients will be collected to the biobank with rheumatoid diseases. These samples will later be used for clinical and basic research, following approval of each specific study by the IRB. The investigators intend to extract protein, DNA and RNA from each sample.

DETAILED DESCRIPTION:
1. PURPOSE Rheumatic diseases, being part of the auto-immune diseases, are rare inflammatory diseases which usually occur from an unknown reason. Various factors alone or in combination can trigger the disease, including pathogens, medications and stress, but the most prominent factor is the genetic background. These diseases are chronic, characterized by periods of flares and regression, and patients are often treated by various drugs. In routine check-up visits in the rheumatology clinic, patients are giving blood regularly in order to monitor the levels of cytokines and antibodies. However, the factors being assessed in the routine lab are limited, and the investigators believe there are much more proteins that can be studied in our research lab. Genomic studies of DNA and RNA isolated from blood of rheumatic patients are rarely being performed, and if they are - only at diagnosis. Combining both protein and genetic profiles of patients at diagnosis and follow up can be extremely useful both for basic and clinical research in helping us to understand the tendency to develop a disease, as well as disease progression and response to therapy. A rheumatoid bio-bank is the basis of establishing many studies leading us a step forward towards personalized medicine.
2. DNA/ RNA resource DNA and RNA will be isolated from blood, synovial fluid or from skin tissue biopsies, related to the rheumatologic disease, derived from patients and normal donors who consent to participate in the rheumatologic Bio-Bank program. The DNA/RNA will be extracted, measured and stored in the bio-bank freezers. Blood samples will be drawn by a physician or accredited nurse, synovial fluid samples and skin biopsies will be collected by physicians only.
3. Patient recruitment: Obtaining Informed Consent

   General Principle:

   Tissues will only be taken from adult patients who gave consent by means of a signed informed consent form.

   All patients above the age of 18, referred to the Rheumatology clinic or Internal Medicine E Department at the Meir Medical Center, for investigation or treatment of suspected rheumatic disease, will be candidates to participate in the repository. Patients at their primary diagnosis or follow up will be eligible for this study. Recruitment of patients and obtaining informed consent will be done by physicians only. No tissue for DNA/RNA isolation will be taken from patients prior to obtaining their written consent or from those who do not consent.

   Number of sample in the bio-bank: 500 for each year
4. Identifying Patients Entitled for Sample Collection 4.1 - General responsibility: The bio bank manager, Dr. Yair Levy, will hold responsibility for appropriate storage and privacy protection of samples, and will be in charge of the bio bank staff.

   4.2- Privacy protection and access to patient's information: To protect patient's privacy identification, a serial code will be generated for each sample. The serial code will replace patient's identifying stickers and along the bio bank processing, samples will only be recognized by bio bank serial codes. The samples are stored in locked freezers or in freezers located in locked rooms accessible to bio bank staff only. The protocol for sample coding: Names and ID numbers of all consented patients will be saved at the bio bank in a separate database that is not connected to the bio bank sample tracking system. On sample reception to the bio bank, the serial code and the correlated patient's identifying number will be recorded on a special secure computer file within the bio bank records. Access to this file will be restricted only to the bio bank coordinator or its manager. All paper documents containing data about patients or samples (e.g. a copy of patients informed consent form) will be kept in locked cabinets.

   4.3 - Coordinating sample collection: The nurse will draw blood according to physician's orders and the attached bio bank forms. Synovial fluid aspirates will be taken solely by physicians and only if medically indicated.

   4.4 - Skin biopsies - The bio bank coordinator will be informed on a weekly basis of all planned skin biopsies at the Dermatology clinic at Meir Medical Center. The biopsy will be performed as clinically needed and with no modification due to banking requirement. All removed tissues will be sent to the pathology lab and processing for banking will begin only after confirmation that adequate tissue is available for the pathology processing. Tissues that eventually will be diagnosed other than rheumatic related disease will be banked and may serve for studies of that specific process or as controls.
5. Participant's rights 5.1 Benefits and risks to participants The impact of human genetics research on human beings is vast. DNA samples taken from patients and volunteers may carry information regarding genetic disorders, inheritance pattern and also about the human nature. The focus of the rheumatologic Bio-bank is on rheumatoid diseases pathogenesis, therapies and immune response during illness and recovery. Samples stored at the Bio-Bank may be subject to any genetic study of rheumatoid diseases regarding the biology, pathogenesis, prognosis, complications or patient's response to the disease or therapy. The benefit outcome from genetic studies to the individual participant may be detection of clinically significant genomic markers which may have implications for patient's appropriate treatment, and follow-up. The risks might include bad mental influence according to one's genetic aberration detected.

   5.2 Withdrawal of participance Participants who want to withdraw their consent must inform the Bio-bank their request in a written letter. Following the acceptance of participant letter, the use of his samples will be immediately stopped and all available DNA samples from this participant will be discarded. In case that a DNA sample from this participant had already been utilized for a specific study, the Bio-bank manager will inform participant request to that study PI which must stop using that sample.

   5.3 Patents rights Participants won't have patent rights or spiritual asset derived from studies that use their samples.

   5.4 Participant's compensation Bio-bank donation will be voluntary only. No compensation will be paid to participants.
6. Timing for Sample Collection and Processing Preferably, the first sample collection should be collected at diagnosis. From patients presented during weekends and holidays the consent will be obtained at admission but samples will be taken early in morning on the first regular working day. It is important that first samples be collected prior to the first drug administration or at least as close to the beginning of therapy as it is possible. By no means will the treatment be delayed for any reason related to this protocol.

Pre-set regular follow-up time points and major clinical events (flare, relapse, and remission) will serve as important milestones. Samples will be drawn simultaneously with the routine clinical tests as ordered by the treating physician. By no means will sample be taken if not otherwise indicated and ordered by the treating physician. All samples should be transported to the laboratory immediately after they had been drawn. Processing should begin as close to the time it was drawn as is possible. Sample Handling protocols 7.1 Sample collection: Blood samples are taken only from participants who have previously consented and authorized the use of their samples for research purposes. Blood will be drawn by any employees certified in taking blood at the Meir Medical Center; synovial fluid will be drawn by physicians only. Blood and synovial fluid will be drawn to lavender and gold top vials with EDTA at a maximum of 20 ml for blood and 30 ml for synovial fluid.

7.2 Blood Processing: Blood samples will be separated to serum and cellular fraction by centrifugation, and kept at -80c until used. White blood cells (WBC) will be collected following red blood cells hemolysis, and stored at -80c. Proteins will be assessed directly from the sera fraction while DNA/RNA will be extracted from WBC.

8. Utilization of frozen sample A. Appreciation for usage of frozen sample

All researchers working at Meir or in any other recognized research institution are potentially eligible for samples use from this protocol. No personal identifying data will be given. A summary of relevant clinical data on the donor of each sample will be enclosed, without any personal data such as name, ID number, hospital record number, address or telephone number. A sample will be eligible for utilization only after the completion of all the following conditions:

1. A written confirmation from the Internal Review Board (IRB) and the head of researcher's institute, approving the specific project / experiment, for which samples are required.
2. The PI of the suggest experiment will present a detailed protocol of the suggested experiment. The protocol should include the rationale and the expected benefit from the experiment, clear and detailed inclusion and exclusion criteria and detailed laboratory protocol.
3. The PI of the suggest experiment will provide a written document listing all samples received for his/her research, confirming his/her obligation and responsibility to follow all ethical roles as detailed by Israeli law and Meir's IRB. The PI of the suggest experiment will not transfer samples to a third party without permission from the Bio-bank manager and the Meir's IRB.
4. The transported samples must be unidentified. Only the Israeli Bio-bank manager will be able to decode the samples information in case it will be needed.
5. The Meir IRB will review all the above documentation and will approve utilizing samples from the Bio Bank.

B. Protocol of tissue usage

Following the completion of all required conditions as mentioned in paragraph A, the PI of the project or experiment should fill out a tissue request form and submit it to the Bio Bank. PI of the Bio Bank project is responsible to verify that all required conditions were fulfilled. The following protocol is to follow:

1. The bio bank coordinator will confirm with the PI who applied for samples when his laboratory team will be ready for picking up samples.
2. Samples will be always dispatched frozen in sealed boxed with dry ice. Samples will be marked with a printed sticker of bio bank barcode of that sample. A detailed summary of the clinical follow up of all patients who donated samples for this project will be attached identified by bio bank barcode only. Names, ID numbers of any other identifying details will not be provided.

C. Utilizing samples priorities and the role for long term banking

1. In case concomitant projects are interested in identical samples: Projects that runs by investigators from Meir Medical Center will be prioritized over projects from other institutes.
2. RNA and DNA will be preferably reserved for large scale studies. International collaborations are welcomed to utilized samples for studies within the scope of this protocol.
3. Samples will be saved as identified samples (as described in 4.2) for 20 years from the end of collection. After 20 years samples will be destroyed unless extending storage duration will approved by Helsinki Committee.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* willing to sign informed consent
* have a rheumatoid condition

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of our rheumatological clinic which have a rheumatolid condition and are willing to sign an informed consent.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2037-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
collecting samples | 20 years
  IgG4-related disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Yair Levy, Prof., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided
we might share samples (serum, DNA, RNA..) but not patient personal details as the samples will be coded.